CLINICAL TRIAL: NCT01969214
Title: Open Label Study to Assess the Safety and Efficacy of IQP-MM-101 in Reducing Symptoms of Diarrhoea
Brief Title: Safety and Efficacy of IQP-MM-101 in Reducing Symptoms of Diarrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INQ/015213
Record Dates: First submitted 2013-10-06; First posted 2013-10-25 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2018-01

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IQP-MM-101 (Experimental): Dissolve the effervescent tablets in half a glass of water,to be taken orally
  1 tablet, 3 times a day
  Interventions: Device: IQP-MM-101

INTERVENTIONS:
Device: IQP-MM-101 — Dissolve the effervescent tablets in half a glass of water, to be taken orally
  1 tablet, 3 times a day

SUMMARY:
Diosmectite in IQP-MM-101 has been used for diarrhoea control. Backed by data from several studies demonstrating their efficacy, the investigators are conducting this study to look into the efficacy and safety of IQP-MM-101 in diarrhoea control.

DETAILED DESCRIPTION:
The clinical study was intended to evaluate the safety and the potential reduction of diarrhoea recovery time post 1st intake of IQP-MM-101 in an open label, single arm, multicentre study over a 72 hours period. There were 2 clinic visits: the screening visit and final visit.

At baseline visit (visit 1), written informed consents were collected. Each patients were given a diary and the following data were collected: demographics, vital signs, physical examination results, use of concomitant medication, previous medical history, and case history of the acute diarrhoea episode including date of first watery stool, number of stools over the past 24 hours, and presence of other associated symptoms over the past 24 hours (nausea, vomiting, abdominal pain).

Subjects recorded the following data in the diary: date and hour of bowel movement, stool consistency (Bristol stool scale) presence of symptoms such as nausea, vomiting, abdominal pain and study IP consumption (number, date, and time of tablets taken) and time of vomiting (if any) each day during the treatment period. Additionally, subjects recorded the time absent from work and a subjective evaluation of their "energy for everyday life".

Visit 2 took place after 72 hours treatment period. Following data was collected:

* Vital signs, physical examination
* Adverse events
* Use of concomitant medication
* Compliance (returned IP and diary)
* Global evaluation of efficacy and safety by subjects and investigators

During the 72-hour treatment period, all subjects were instructed to consumed IQP-MM-101 according to the following dosage: one (1) tablet, three (3) times a day dissolved in at least 125mL (half a glass) of water.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Good general health
* Acute diarrhoea episode defined as at least three watery stools per 24 hours over a period of 48 hours or less
* Acute diarrhoea of presumed infectious origin
* Patients with usually normal bowel movements (defecations) before onset of diarrhoea, that is, at least three normal stools per week and three or less normal stools per day
* Negative pregnancy test (ß HCG-test) for women with child bearing potential
* Written informed consent is a prerequisite for subject enrollment

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Fever >38,5◦C
* Blood or pus in stools
* Dehydration requiring intravenous rehydration
* History of chronic diarrhoea (three or more loose or watery stools per day for at least 12 weeks, consecutive or not, in the preceding 12 months)
* Use of antidiarrhoeal agents over the month prior to baseline
* Diarrhoea possibly induced by antibiotics, laxative agents, thyroid hormones, or colchicine
* Irritable bowel syndrome
* Any other acute or chronic disease that could interfere with the evaluation of study device
* Females who are pregnant or lactating
* Subjects who have participated in another clinical trial in the 30 days before treatment period
* Inability to comply
* Presence of other factor(s) that, in the investigator's judgement, should preclude subject participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IQP-MM-101: Dissolve the effervescent tablets in half a glass of water,to be taken orally
  1 tablet, 3 times a day
  IQP-MM-101: Dissolve the effervescent tablets in half a glass of water, to be taken orally
  1 tablet, 3 times a day
Period: Overall Study
Arm/Group | IQP-MM-101
Started | 101
Completed | 86
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population consisted of all subjects who received at least one dose of investigational product (intent to treat). In cases where all dispensed investigational product is returned, the subject was considered non-treated and therefore was not included in the FAS.
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (11.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 46
Region of Enrollment [Number; unit: participants]
  Germany | 86

OUTCOME MEASURES:

1. Primary Outcome: Time (in Hours) Between the 1st Intake of IQP-MM-101 and First Formed or Hard Stool (Type 6 to 1) Followed by a Non Watery Stool (Type 6 to 1)
Description: In essence the definition of recovery would be two consecutive non-watery stool (type 6 to 1) when stool before 1st intake of IQP-MM-101 is primarily watery (type 7).
Time Frame: 96 hours
Population: 6 participants recovered before first intake of IQP-MM-101, while in another, there was no defecation reported.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 79
hours | 21.30 (16.02)

2. Secondary Outcome: Time (Hours) From the First Intake to the Last Watery Stool
Description: The last watery stool was assumed as the first-non watery stool
Time Frame: 96 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 79
Hours | 18.17 (15.85)

3. Secondary Outcome: Number of Daily Defecation
Time Frame: 96 hours
Measure: Number; unit: stools
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
stools
  Day 1 | 387
  Day 2 | 278
  Day 3 | 200
  Day 4 | 82

4. Secondary Outcome: Number of Watery Stools
Time Frame: 96 hours
Measure: Number; unit: stools
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
stools
  Day 1 | 292
  Day 2 | 72
  Day 3 | 20
  Day 4 | 10

5. Secondary Outcome: Stool Frequency
Description: The mean number of daily defecation.
Time Frame: 96 hours
Measure: Mean (Standard Deviation); unit: No. of daily defecation
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
No. of daily defecation
  Stool Frequency Day 1 | 4.50 (2.57)
  Stool Frequency Day 2 | 3.23 (1.90)
  Stool Frequency Day 3 | 2.33 (1.58)
  Stool Frequency Day 4 | 0.95 (1.03)

6. Secondary Outcome: Percentage of Patients Having Recovered Within a Certain Time Period (Defined as Having Achieved the Primary Efficacy Endpoint)
Time Frame: 72 hours
Measure: Number; unit: Percentage of subjects
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 79
Percentage of subjects
  Recovery time: Up to 24 hours | 25.3
  Recovery time: More than 24 up to 30 hours | 21.5
  Recovery time: More than 30 up to 36 hours | 8.9
  Recovery time: More than 36 up to 42 hours | 7.6
  Recovery time: More than 42 up to 48 hours | 16.5
  Recovery time: More than 48 up to 60 hours | 10.1
  Recovery time: More than 60 up to 72 hours | 8.9
  Recovery time: More than 72 hours | 1.3

7. Secondary Outcome: Abdominal Pain
Description: Subjects feeling of abdominal pain was measured on visual analog scale of 0 - 100mm (no pain to severe pain).
Time Frame: 96 hours
Population: All 86 subjects recorded abdominal pain on day 1 and day 2. 85 subjects recorded abdominal pain on day 3 and 67 subjects recorded abdominal pain on day 4.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
mm
  Severity of abdominal pain Day 1 | 56.2 (23.6)
  Severity of abdominal pain Day 2 | 35.3 (20.8)
  Severity of abdominal pain Day 3: number analyzed (Participants) | 85
  Severity of abdominal pain Day 3 | 18.7 (16.7)
  Severity of abdominal pain Day 4: number analyzed (Participants) | 67
  Severity of abdominal pain Day 4 | 11.1 (14.3)

8. Secondary Outcome: Time Off From Work
Time Frame: 1 week
Measure: Number; unit: Percentage of subjects
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
Percentage of subjects
  0 day of absent | 31.4
  1 day of absent | 4.7
  2 days of absent | 11.6
  3 days of absent | 7.0
  4 days of absent | 12.8
  5 days of absent | 24.4
  More than 6 days of absent | 8.1

9. Secondary Outcome: Evaluation of Subjects' Energy Level
Description: The subjective measure of subjects' daily energy level was determined by severity of weakness felt by the subjects, measured on visual analog scale (0-100mm, 100mm being most severe weakness).
Time Frame: 96 hours
Population: Only 85 subjects responded to Day 3 and only 67 subjects responded to Day 4 assessment of weakness
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
mm
  Severity of Weakness Day 1 | 67.5 (21.5)
  Severity of Weakness Day 2 | 45.7 (24.7)
  Severity of Weakness Day 3: number analyzed (Participants) | 85
  Severity of Weakness Day 3 | 29.5 (24.6)
  Severity of Weakness Day 4: number analyzed (Participants) | 67
  Severity of Weakness Day 4 | 16.8 (19.7)

10. Secondary Outcome: Global Evaluation of Safety and Efficacy by Subjects and Investigators
Description: The subjects and investigators will evaluate independently the safety of the investigational device (global scaled evaluation with "very good", "good", "moderate" and "poor").
Time Frame: 96 hours
Measure: Number; unit: participants
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
participants
  Efficacy by Investigator - Very Good | 21
  Efficacy by Investigator - Good | 61
  Efficacy by Investigator - Moderate | 2
  Efficacy by Investigator - Poor | 2
  Efficacy by Subjects - Very Good | 28
  Efficacy by Subjects - Good | 54
  Efficacy by Subjects - Moderate | 2
  Efficacy by Subjects - Poor | 2
  Safety by Investigator - Very Good | 51
  Safety by Investigator - Good | 34
  Safety by Investigator - Moderate | 1
  Safety by Investigator - Poor | 0
  Safety by Subjects - Very Good | 50
  Safety by Subjects - Good | 36
  Safety by Subjects - Moderate | 0
  Safety by Subjects - Poor | 0

11. Secondary Outcome: Occurrence of Adverse Events (AEs)
Time Frame: 96 hours
Measure: Number; unit: Adverse Events
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 99
Adverse Events | 7

12. Secondary Outcome: Associated Symptoms Such as Vomiting
Time Frame: 96 hours
Measure: Number; unit: Percentage of subjects
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
Percentage of subjects
  Affected subjects at day 1 | 23.3
  Affected subjects at day 2 | 3.5
  Affected subjects at day 3 | 3.5
  Affected subjects at day 4 | 3.5

13. Secondary Outcome: Stool Consistency
Description: Stool consistency is measured by Bristol Stool Form Scale 1-7.
  1. Separate hard lumps, like nuts (hard to pass)
  2. Sausage-shaped, but lumpy
  3. Like a sausage but with cracks on its surface
  4. Like a sausage or snake, smooth and soft
  5. Soft blobs with clear cut edges (easy to pass)
  6. Fluffy pieces with ragged edges, a mushy stool
  7. Watery, no solid pieces, entirely liquid Stool consistency is the mean of the scale measured each day.
Time Frame: 96 hours
Population: 387, 278, 200 and 82 stool samples were obtained on day 1, 2, 3 and 4 respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: stool samples
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
Number analyzed (stool samples) | 387
score on a scale
  Type of Stool Day 1 | 6.66 (0.84)
  Type of Stool Day 2: number analyzed (stool samples) | 278
  Type of Stool Day 2 | 5.83 (1.33)
  Type of Stool Day 3: number analyzed (stool samples) | 200
  Type of Stool Day 3 | 4.18 (1.50)
  Type of Stool Day 4: number analyzed (stool samples) | 82
  Type of Stool Day 4 | 3.32 (1.25)

14. Secondary Outcome: Severity of Nausea
Description: Subjects feeling of nausea was measured on visual analog scale of 0 - 100mm (no nausea to severe nausea).
Time Frame: 96 hours
Population: All 86 subjects recorded nausea on day 1 and day 2. 85 subjects recorded nausea on day 3 and 67 subjects recorded nausea on day 4.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IQP-MM-101
Number analyzed (Participants) | 86
mm
  Severity of nausea Day 1 | 44.8 (29.5)
  Severity of nausea Day 2 | 28.1 (23.4)
  Severity of nausea Day 3: number analyzed (Participants) | 85
  Severity of nausea Day 3 | 12.9 (16.0)
  Severity of nausea Day 4: number analyzed (Participants) | 67
  Severity of nausea Day 4 | 8.3 (13.7)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | IQP-MM-101
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 6/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQP-MM-101 (N=99)
Cold (General disorders) | 2 (2)
Cough (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Tinea Corporis (Infections and infestations) | 1 (1)
Heartburn (General disorders) | 1 (1)
Viral Infection of the Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No